CLINICAL TRIAL: NCT07049250
Title: Effect of Evidence-Based Nursing Intervention Under Quantitative Evaluation Strategy on Psychological Resilience and Illness Perception in Lung Cancer Patients Undergoing Chemotherapy
Brief Title: Evidence-Based Nursing for Psychological Resilience in Lung Cancer Chemotherapy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Feifei Wang, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024S00040
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: Chemotherapy; Psychological Resilience; Illness Perception; Evidence-Based Nursing; Quantitative Evaluation Strategy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-Based Nursing Intervention Group (Experimental): Participants (n=71) received evidence-based nursing intervention guided by quantitative evaluation strategy. This included: 1) comprehensive risk assessments by a multidisciplinary team; 2) dynamic risk stratification for care intensity; 3) psychological and cognitive interventions (cognitive-behavioral techniques, peer mentoring, family counseling); 4) systematic complication prevention strategies (prophylactic antiemetics, dietary guidance, infection control); 5) sleep optimization protocols.
  Interventions: Behavioral: Evidence-Based Nursing Intervention under Quantitative Evaluation Strategy
- Routine Nursing Care Group (Active Comparator): Participants (n=71) received routine nursing care. This consisted of standard disease education covering chemotherapy side effects and self-management strategies, personalized exercise guidance focusing on maintaining physical function, and medication adherence counseling, delivered in 30-minute sessions twice weekly for a duration of two months.
  Interventions: Behavioral: Routine Nursing Care

INTERVENTIONS:
Behavioral: Evidence-Based Nursing Intervention under Quantitative Evaluation Strategy — A multifaceted nursing program incorporating comprehensive risk assessment, dynamic risk stratification, psychological and cognitive interventions (including cognitive-behavioral techniques, peer mentoring, family counseling), systematic complication prevention strategies (including prophylactic antiemetics, dietary guidance, infection control), and sleep optimization protocols.
  Arms: Evidence-Based Nursing Intervention Group
Behavioral: Routine Nursing Care — Standard disease education on chemotherapy side effects and self-management, personalized exercise guidance, and medication adherence counseling. Delivered in 30-minute sessions twice weekly for two months.
  Arms: Routine Nursing Care Group

SUMMARY:
This study investigates the effect of an evidence-based nursing intervention, guided by a quantitative evaluation strategy, on psychological resilience and illness perception in lung cancer patients undergoing chemotherapy. Patients were randomized to receive either the specialized nursing intervention or routine nursing care, with outcomes assessed at baseline and 3 months post-intervention.

DETAILED DESCRIPTION:
Lung cancer patients undergoing chemotherapy often experience significant physical and psychological distress. Conventional nursing may not adequately address these multifaceted needs. Evidence-based nursing (EBN) integrates research evidence, clinical expertise, and patient preferences. This study evaluated an EBN intervention model guided by a quantitative evaluation strategy, which involves multidisciplinary risk assessment, tailored interventions including psychological support, cognitive restructuring, and complication prevention. The study aimed to determine if this model could improve psychological resilience, illness perception, coping styles, and reduce chemotherapy-related complications in lung cancer patients compared to routine nursing care. A total of 142 patients were randomized. The intervention group received a comprehensive EBN program including risk stratification, psychological/cognitive interventions (e.g., cognitive-behavioral techniques, peer mentoring, family counseling), systematic complication prevention (e.g., prophylactic antiemetics, dietary guidance, infection control), and sleep optimization. The control group received standard disease education, exercise guidance, and medication adherence counseling. Outcomes were measured at baseline and 3 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung cancer confirmed according to the Chinese Quality Control Indicators for Standardized Diagnosis and Treatment of Primary Lung Cancer (2022) through both imaging and histopathological examination.
* TNM staging determined using the 8th edition AJCC/UICC classification system.
* Scheduled to receive chemotherapy with an expected survival exceeding one year.
* Demonstrated normal cognitive and communication abilities as assessed by standardized neuropsychological tests.
* Provided written informed consent prior to enrollment.

Exclusion Criteria:

* Pre-existing neurological disorders.
* Significant organ dysfunction (defined as Child-Pugh class B/C for liver function or eGFR <30 mL/min/1.73m² for renal function).
* Active infectious diseases.
* Contraindications to chemotherapy.
* Concurrent radiotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Resilience Score | Baseline and 3 months post-intervention.
  Psychological resilience assessed using the 25-item Resilience Scale. Scores range from 0 to 100, with higher scores indicating better psychological resilience. The scale measures optimism, resilience, and strength subdomains.

SECONDARY OUTCOMES:
Change in Illness Perception | Baseline and 3 months post-intervention.
  Illness perception assessed using the Brief Illness Perception Questionnaire (B-IPQ). This evaluates emotional, cognitive, and comprehension domains, with each item scored from 0 to 10. Higher scores in relevant domains indicate more positive or accurate illness perception.
Change in Coping Styles | Baseline and 3 months post-intervention.
  Coping styles measured by the Simplified Coping Style Questionnaire (SCSQ) to distinguish between active and passive coping strategies. Higher scores for active coping and lower scores for passive coping are generally considered favorable.
Incidence of Chemotherapy-Related Complications | Assessed throughout the 3-month post-intervention period.
  Occurrence of chemotherapy-related complications including gastrointestinal reactions, pulmonary infections, hepatorenal toxicity, bone marrow suppression, and phlebitis. Assessed as percentage of patients experiencing each complication.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China